CLINICAL TRIAL: NCT06271707
Title: Left Sided Stellate Ganglion Blocks Impact on the Rate of Post-operative Atrial Fibrillation in Patients Undergoing Thoracic Surgery: A Pilot Study
Brief Title: Stellate Ganglion Block
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ANES-2024-32720
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Esophagectomy; Pneumonectomy; Lobectomy
Keywords: Esophagectomy; Pneumonectomy; Lobectomy; Stellate Ganglion Block
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double blind randomized prospective controlled trial. Randomization will be 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): ultrasound with bupivacaine
  Interventions: Drug: 0.5% bupivacaine
- Group 2 (Sham Comparator): Ultrasound with saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: 0.5% bupivacaine — an ultrasound guided left stellate ganglion block with 5 mL of 0.5% bupivacaine
  Arms: Group 1
Other: Saline — an ultrasound guided left stellate ganglion block with 5 mL of saline
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine if the addition of an ultrasound guided left sided stellate ganglion block with bupivacaine in patients undergoing esophagectomy, pneumonectomy, or lobectomy will result in lower rates of postoperative atrial fibrillation as compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophagectomy, pneumonectomy, or lobectomy aged 18-85.

Exclusion Criteria:

* Patients who have an exclusion to regional anesthesia.
* Patients who have exclusion to stellate blockade.
* Patients who are pregnant assessed via self-report or pregnancy test if they have taken one

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
an ultrasound guided left stellate ganglion block with 5 mL of saline. | 168 hours after surgery
  Incidence of Atrial fibrillation in the first 168 hours after surgery.
Atrial fibrillation; Other arrhythmias; Adverse events. | 168 hours after surgery
  Atrial fibrillation in first 24, 48, 72, 96, 120, and 144 hours; Other arrhythmias in first 24, 48, 72, 96, 120, 144 and 168 hours; Adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hutchins, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States